CLINICAL TRIAL: NCT00003982
Title: Phase I Study to Determine the Safety of MEN-10755 (BMS-195615) in Patients With a Solid Tumor on a Short I.V. Infusion Given Once Every Week for 3 Consecutive Weeks, Followed by One Week's Rest
Brief Title: MEN-10755 in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16970; EORTC-16970
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; testicular embryonal carcinoma and yolk sac tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Endodermal Sinus Tumor | interventions — sabarubicin

INTERVENTIONS:
Drug: sabarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of MEN-10755 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of MEN-10755 in patients with solid tumors. II. Determine the qualitative and quantitative toxic effects of this drug and study the predictability, duration, intensity, onset, reversibility and dose relationship of the toxic effects in this patient population. III. Propose a safe dose for phase II study. IV. Study the pharmacokinetics of this drug at different dose levels in this patient population. V. Document any possible antitumor activity of this drug in this patient population.

OUTLINE: This is a dose escalation study. Patients receive MEN-10755 IV over 15 minutes on days 1, 8, and 15. Treatment continues every 4 weeks, or upon recovery of toxicity, whichever comes later. Treatment continues for at least 2 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of MEN-10755 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed for at least 3 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor that is not amenable to standard therapy Measurable or evaluable disease No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Liver function tests no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.4 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: LVEF at least 50% (by MUGA) Other: Not pregnant or nursing Fertile patients must use effective contraception No active infections No other nonmalignant disease that precludes study No history of alcoholism, drug addiction, or psychotic disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, and high dose carboplatin) No other concurrent antitumor drugs Endocrine therapy: No concurrent corticosteroids Radiotherapy: At least 4 weeks since prior radiotherapy (6 weeks for extensive radiotherapy) No concurrent radiotherapy Surgery: Not specified Other: No prior anthracyclines or anthracenediones No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: Emma Geertruida Elisabeth De Vries, MD, PhD, Study Chair — University Medical Center Groningen
Locations (27):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland